CLINICAL TRIAL: NCT03121378
Title: Multiple Electrode Aggregometry to Assess Platelet Function in Patients Undergoing Hip Joint Alloplasty With and Without Bone Cement
Acronym: APJAB
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marek Janiak, Dr, Medical University of Warsaw
Other Study IDs: APJAB
Record Dates: First submitted 2017-04-12; First posted 2017-04-20 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Arthroplasty; Methylmethacrylate Embolism; Platelet Aggregation
Keywords: Hip Joint Alloplasty; Bone Cements; Impedance Aggregometry; Platelet Activation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3ml Blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hip arthroplasty with bone cement: Patients undergoing hip replacement surgery with bone cement use: blood samples taken before cement use and after cement prosthesis fixation.
  Interventions: Other: Blood sample 1; Other: Blood sample 2
- Non cement hip arthroplasty: Patients undergoing hip replacement surgery without bone cement. Blood samples taken before bone reaming and after implantation of femoral prosthesis.
  Interventions: Other: Blood sample 1; Other: Blood sample 2

INTERVENTIONS:
Other: Blood sample 1 — Blood taken before prosthesis implantation
Other: Blood sample 2 — Blood taken after prosthesis implantation

SUMMARY:
The aim of the study is to assess blood platelet function and activation in patients undergoing both cement and non cement hip joint total alloplasty. Bone cement is used as a special biomaterial to help fix a hip prosthesis in place but is associated with bone cement implantation syndrome causing such complications as hypotension, cardiac arrhythmias. The pathophysiology of bone cement implantation syndrome is not fully known but one theory supports formation of clots in the bloodstream. This directly would activate platelets but no such study has been performed in humans. As bone reaming could potentially cause platelet activation even without bone cement, the study involves a control group of patients undergoing non cemented joint alloplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients qualified for hip arthroplasty
* Signed consent for study
* No abnormality in coagulation screen
* Not taking regular antiplatelet medication except small dose of acetylsalicylic acid

Exclusion Criteria:

* Lack of consent
* Low platelet count (<100 thousand) in standard preoperative full blood count
* On regular antiplatelet medication (except 75mg acetylsalicylic acid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing hip arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Change in platelet aggregation as expressed by height and slope of curve | Up to 30 minutes
  Differences in increase of impedance to a current during multiple electrode aggregometry measured as area under curve (AUC) expressed in units AU*minute which is derived from the velocity and maximum height of the aggregometry curves

CONTACTS AND LOCATIONS:
Locations (1):
- I Department of Anesthesiology and Intensive Care Warsaw Medical University, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No